CLINICAL TRIAL: NCT04089748
Title: Basal Tumours in Bladder Cancer, Response to chemoTherapy
Acronym: BoBCaT
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut Curie (Other); APHP (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/384/HP
Record Dates: First submitted 2019-09-04; First posted 2019-09-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Bladder Cancer; Chemotherapy Effect
Keywords: neoadjuvant chemotherapy; cisplatine
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients enrolled in VESPER study: Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in VESPER cohort
  Interventions: Combination Product: neoadjuvant chemotherapy with cisplatine
- Patients from St Louis cohort not enrolled in VESPER study: Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in Saint-Louis cohort
  Interventions: Combination Product: neoadjuvant chemotherapy with cisplatine

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy with cisplatine — Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine

SUMMARY:
Determine the sensitivity/resistance to chemotherapy of the various subgroups of muscle-invasive bladder cancers, including the basal subgroup (about 25% of these tumours) according to 4 different classifications based on molecular or immunohistochemical classifiers.

ELIGIBILITY:
Inclusion Criteria of Patients enrolled in VESPER study:

Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in VESPER cohort and :

* having signed an informed consent form for the participation to the collection or
* dead/lost to follow-up without prior opposition expressed against research program,
* genetic analysis will only be carried out for patients who have signed the genetic consent form.

Inclusion Criteria of Patients from St Louis cohort not enrolled in VESPER study:

Tumors from patient having muscle invasive bladder cancer who benefit from neoadjuvant chemotherapy with cisplatine included in Saint-Louis cohort and :

* having received an informed form for the participation to the collection and not having expressed opposition against research program within 1 month or
* dead/lost to follow-up without prior opposition expressed against research program,

Exclusion Criteria:

-Patients enrolled in VESPER study:Tumors from patient having withdrawn his/her informed consent form for the participation to the collection and/or VESPER project.

OR

-Patients from St Louis not enrolled in VESPER study:Tumors from patient having expressed opposition against research program after 1 month for the participation to the collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumors from patient having muscle invasive bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Identifying molecular subgroups of bladder cancer patients within VESPER and Saint-Louis cohort, who could benefit from neoadjuvant chemotherapy, taking into account the existence of different classification systems. | through study completion, an average of 3 years
Determining which classification(s) has(ve) the best ability to identifying subgroups of tumours sensitive or resistant to neoadjuvant chemotherapy. | through study completion, an average of 3 years
Identifying mechanisms of resistance in basal subgroups. | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- DRCI, Rouen, France

IPD SHARING:
Plan to Share IPD: No